CLINICAL TRIAL: NCT02612870
Title: Sienna+® Injection Time Study: A Prospective Multicentre, Controlled Clinical Trial to Evaluate the Performance of Superparamagnetic Iron Oxide vs. Standard Technique as Tracer in Sentinel Node Biopsy
Brief Title: Sienna+® Injection Time Study 4 Arms
Acronym: Sentimag02
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kantonsspital Baden (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Principal Investigator, Nik Hauser, Director Department of Gynecology and Obstetrics, Kantonsspital Baden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Baden201512
Record Dates: First submitted 2015-11-18; First posted 2015-11-24 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: Breast Neoplasms
Keywords: Breast Cancer; Sentinel Node; Sentinel Node Biopsy; Breast Surgery
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sienna+ retro and Technetium 1 (Active Comparator): Sienna+® is administered retro-mamillary 1 day before surgery for sentinel node marking.
  Technetium as standard technique is employed according to the gold standard protocol one day before surgery.
  The Sentimag device is used during surgery to detect the lymph nodes in parallel to the standard technique.
  Interventions: Device: Sienna+ retro; Device: Technetium 1
- Sienna+ peri and Technetium 1 (Active Comparator): Sienna+® is administered peri-tumorally 1 day before surgery for sentinel node marking.
  Technetium as standard technique is employed according to the gold standard protocol one day before surgery.
  The Sentimag device is used during surgery to detect the lymph nodes in parallel to the standard technique.
  Interventions: Device: Sienna+ peri; Device: Technetium 1
- Sienna+ retro 4-6 and Technetium 1 (Active Comparator): Sienna+® is administered retro-mamillary 4-6 days before surgery for sentinel node marking.
  Technetium as standard technique is employed according to the gold standard protocol one day before surgery.
  The Sentimag device is used during surgery to detect the lymph nodes in parallel to the standard technique.
  Interventions: Device: Sienna+ retro 4-6; Device: Technetium 1
- Sienna+ peri 4-6 and Technetium 1 (Active Comparator): Sienna+® is administered peri-tumorally 4-6 days before surgery for sentinel node marking.
  Technetium as standard technique is employed according to the gold standard protocol one day before surgery.
  The Sentimag device is used during surgery to detect the lymph nodes in parallel to the standard technique.
  Interventions: Device: Sienna+ peri 4-6; Device: Technetium 1

INTERVENTIONS:
Device: Sienna+ retro — Sentinel node marking with Sienna+ retro-mamillary 1 day before surgery
  Arms: Sienna+ retro and Technetium 1
Device: Sienna+ peri — Sentinel node marking with Sienna+ peri-tumorally 1 day before surgery
  Arms: Sienna+ peri and Technetium 1
Device: Sienna+ retro 4-6 — Sentinel node marking with Sienna+ retro-mamillary 4-6 days before surgery
  Arms: Sienna+ retro 4-6 and Technetium 1
Device: Sienna+ peri 4-6 — Sentinel node marking with Sienna+ peri-tumorally 4-6 days before surgery
  Arms: Sienna+ peri 4-6 and Technetium 1
Device: Technetium 1 — Sentinel node marking with Technetium 1 day before surgery

SUMMARY:
Patients with breast cancer normally undergo a labelling with radioactive tracer typically 1 day before surgery, which enables the surgeon to localize the sentinel lymph node during surgery. This pilot study uses the magnetic Sentimag technique to mark the lymph nodes either 1 or 4-6 days before surgery to investigate the concordance with the standard technique.

DETAILED DESCRIPTION:
Sienna+® is injected either 1 day or 4-6 days before surgery, either retro-mamillary or peri-tumorally:

* Sienna+® retro-mamillary 1 day before surgery: 10 patients
* Sienna+® peri-tumorally 1 day before surgery: 10 patients
* Sienna+® retro-mamillary 4-6 days before surgery: 10 patients
* Sienna+® peri-tumorally 4-6 days before surgery: 10 patients In each case, Technetium as standard technique is employed according to the gold standard protocol one day before surgery.

The Sentimag device is used during surgery to detect the lymph nodes in parallel to the standard technique.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a diagnosis of primary breast cancer
* Subject has been scheduled for surgery with a sentinel lymph node biopsy procedure
* Subject is ≥18 years old at time of consent
* Subject has an ECOG performance status of Grade 0-2
* Subject has a clinical negative node status
* Subject is available for the follow-up

Exclusion Criteria:

* Subject is pregnant or lactating
* Subject has a radiological evidence of metastatic cancer
* Subject has had previous axilla surgery or reduction mammoplasty
* Subject has impaired lymphatic function
* Subject has had a preoperative radiation therapy
* Subject has iron overload disease or iron/dextran intolerance
* Subject has a pacemaker
* Subject is under guardianship

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Detection rate per Patient | During surgery
  Proportion of successfully detected sentinel nodes (detection rate per patient) with both methods.

SECONDARY OUTCOMES:
Number of lymph nodes excised | During surgery
  Number of excised sentinel lymph nodes
Nodal detection rate | During surgery
  Number of detected versus excised sentinel lymph nodes with either method.
Malignancy rate | 1-2 days post surgery
  Number of histologically confirmed malignant sentinel lymph nodes detected with either method.

CONTACTS AND LOCATIONS:
Overall Officials: Nik Hauser, PD Dr., Principal Investigator — Kantonsspital Baden
Locations (2):
- Switzerland (2):
  - Kantonsspital Baden, Baden
  - Inselspital Bern, Universitätsklinik für Frauen., Bern

REFERENCES:
- [Result] Thill M, Kurylcio A, Welter R, van Haasteren V, Grosse B, Berclaz G, Polkowski W, Hauser N. The Central-European SentiMag study: sentinel lymph node biopsy with superparamagnetic iron oxide (SPIO) vs. radioisotope. Breast. 2014 Apr;23(2):175-9. doi: 10.1016/j.breast.2014.01.004. Epub 2014 Jan 29. PMID 24484967
- [Result] Douek M, Klaase J, Monypenny I, Kothari A, Zechmeister K, Brown D, Wyld L, Drew P, Garmo H, Agbaje O, Pankhurst Q, Anninga B, Grootendorst M, Ten Haken B, Hall-Craggs MA, Purushotham A, Pinder S; SentiMAG Trialists Group. Sentinel node biopsy using a magnetic tracer versus standard technique: the SentiMAG Multicentre Trial. Ann Surg Oncol. 2014 Apr;21(4):1237-45. doi: 10.1245/s10434-013-3379-6. Epub 2013 Dec 10. PMID 24322530
- [Result] Ghilli M, Carretta E, Di Filippo F, Battaglia C, Fustaino L, Galanou I, Di Filippo S, Rucci P, Fantini MP, Roncella M. The superparamagnetic iron oxide tracer: a valid alternative in sentinel node biopsy for breast cancer treatment. Eur J Cancer Care (Engl). 2017 Jul;26(4). doi: 10.1111/ecc.12385. Epub 2015 Sep 14. PMID 26365441
- [Result] Rubio IT, Diaz-Botero S, Esgueva A, Rodriguez R, Cortadellas T, Cordoba O, Espinosa-Bravo M. The superparamagnetic iron oxide is equivalent to the Tc99 radiotracer method for identifying the sentinel lymph node in breast cancer. Eur J Surg Oncol. 2015 Jan;41(1):46-51. doi: 10.1016/j.ejso.2014.11.006. Epub 2014 Nov 15. PMID 25466980